CLINICAL TRIAL: NCT06634160
Title: Assessment of Metabolic Dysfunction-associated Steatotic Liver Disease (MASLD) Prevalence in Patients With Heterozygous Familial Hypercholesterolemia (HeFH): the STEATO-FH Study
Brief Title: Assessment of the Prevalence of Steatotic Liver Disease Associated With Metabolic Dysfunction in Patients With Heterozygous Familial Hypercholesterolemia
Acronym: STEATO-FH
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: University Hospital, Angers (Other Government); Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC24_0064; 2024-A01647-40 (Other: IDRCB (ANSM))
Record Dates: First submitted 2024-10-04; First posted 2024-10-09 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Heterozygous Familial Hypercholesterolemia
Keywords: MASLD; Heterozygous Familial Hypercholesterolemia; steatosis; fibrosis
MeSH Terms: conditions — Fatty Liver; Fibrosis | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Two tubes of 10 mL blood each will be collected per patient in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study population: The study population must correspond to the research inclusion criteria. A fibroscan will be performed on each patient enrolled in the study. Each participant will also be offered a biological sample for an ancillary study.
  Interventions: Diagnostic Test: Fibroscan; Other: Sample collection

INTERVENTIONS:
Diagnostic Test: Fibroscan — Evaluation of the prevalence of steatosis by measuring ultrasound attenuation with Fibroscan® (non-invasive method, at a distance from a meal (3h fasting)).
Other: Sample collection — 20 mL whole blood sample

SUMMARY:
The main goal of the STEATO-FH study is to determine the prevalence of liver steatosis within the Heterozygous Familial Hypercholesterolemia patient population.

DETAILED DESCRIPTION:
Investigators will include patients being followed for heterozygous familial hypercholesterolemia in their centers. The prevalence of hepatic steatosis will be studied non-invasively, using Fibroscan ®. In addition, coronary calcium score (CAC scores) will be evaluated and a biocollection will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 35 or over
* Consultation at Nantes, Rennes or Angers University Hospital during the inclusion period
* With a diagnosis of familial hypercholesterolemia defined by the presence of a genetic variant, ACMG classes 4 & 5 on LDLR, APOB or PCSK9
* Patient not objecting to inclusion in study (no written objection)

Exclusion Criteria:

* Protected patients: minors, adults under guardianship, curatorship and/or safeguard of justice
* Pregnant or breast-feeding
* Active viral hepatitis
* Hemochromatosis
* Other genetic or autoimmune hepatitis
* Current treatment with a drug likely to cause hepatic steatosis, including amiodarone, carbamazepine, tamoxifen, valproate, clozapine, anti-retrovirals
* Current oral corticosteroid therapy unless dose has been stable for ≥ 3 months
* Current pathological alcohol consumption (≥ 60 g/day in men and ≥ 50 g/day in women)

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients are those with definite familial hypercholesterolemia (genetic variant, ACMG classes 4 & 5 on LDLR, APOB or PCSK9), consulting during the inclusion period and age ≥ 35 years.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Presence of steatosis in HeFH patients | 1 day
  Presence of steatosis in HeFH patients assessed by Fibroscan® measurement of CAP (Controlled Attenuation Parameter) ≥ 275 dB/m (Berzigotti et al., 2021)

SECONDARY OUTCOMES:
Establish the prevalence of hepatic fibrosis | 1 day
Evaluate the prevalence of diabetes among HeFH patients, according to the presence or absence of steatosis or fibrosis | 1 day
Evaluate the association between anthropometric measures (weight, height, waist circumference, and calculated BMI) and the presence of hepatic steatosis or fibrosis. | 1 day
Evaluate the association between LDL-cholesterol and time of exposure to elevated LDL-cholesterol (Gallo et al. J Clin Lipidol 2017) with the prevalence of steatosis or fibrosis | 1 day
Evaluate the proportion of patients with hepatic steatosis or fibrosis according to the nature of the genetic mutation | 1 day
Evaluate the link between the presence of hepatic steatosis or fibrosis and the risk of cardiovascular disease | 12 months
Determine factors associated with the presence of steatosis or hepatic fibrosis | 1 day

OTHER OUTCOMES:
Identify blood biomarkers associated with hepatic steatosis and fibrosis | 1 day

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU angers, Angers
  - CHU Nantes, Nantes
  - Rennes University Hospital, Rennes